CLINICAL TRIAL: NCT01458678
Title: Evaluation of Non Invasive Methods for Goal Directed Fluid Therapy During Abdominal Surgery
Brief Title: Non Invasive Methods to Guide Volume Optimization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lena Nilsson (Other)
Responsible Party: Sponsor-Investigator, Lena Nilsson, Senior consultant, PhD, University Hospital, Linkoeping
Organization: University Hospital, Linkoeping (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PVI vers OD
Record Dates: First submitted 2011-10-20; First posted 2011-10-25 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oesophageal Doppler (OD) (Active Comparator): Goal directed volume therapy is most often guided by stroke volume measurements by OD.
  Interventions: Other: Volume of colloid infusion
- Pleth Variability Index (PVI) (Active Comparator): The Pleth variability index (PVI) is an automated function in pulse oximetry that continuously calculates the dynamic variation between the pulse oximetry pulse variation and its baseline for every breathing circuit. Dynamic indicators are advantageous in predicting a responder to a volume bolus, thus facilitating goal directed volume therapy.
  Interventions: Other: Volume of colloid infusion

INTERVENTIONS:
Other: Volume of colloid infusion — Colloid infusion is primarily given as hydroxyethyl starch 60 mg/ml. If more than 30 ml/kg hydroxyethyl starch 60 mg/ml is given, colloid solution is changed to albumin 4% or plasma.
  Arms: Oesophageal Doppler (OD)
Other: Volume of colloid infusion — Colloid infusion is given primarily as hydroxyethyl starch 60 mg/ml. If more than 30 ml/kg hydroxyethyl starch 60 mg/ml is given, colloid solution is changed to albumin 4% or plasma.
  Arms: Pleth Variability Index (PVI)

SUMMARY:
Goal directed volume therapy means that bolus doses of 150-250 ml colloid fluid is administered to the patient during contemporary measurement of the patients stroke volume. The fluid status is considered optimized when stroke volume no longer increases with more than 10%, indicating that the patient is close to the top of the Frank-Starling curve. Several studies show that volume optimization reduces hospital stay and reduces the amount of surgical complications. The overall purpose is to investigate if the much more simple non invasive technique Pleth Variability Index can replace oesophageal doppler to guide volume therapy in routine health care, and to analyse if a volume kinetic test can be used to evaluate hypovolemia before surgery and make specific rehydration possible by analysing the correlation between this test and fluid optimization using stroke volume measurements.

Primary hypothesis: 1. The volume of colloids that is given to volume optimise an anesthetized patient using Pleth Variability Index shows a good correlation to the volume used if volume optimisation is undertaken by the guidance of oesophageal doppler. 2. Data from the two methods correlate and discriminates similarly volume responders from non responders. 3. A volume kinetic model that indicates dehydration can predict the need for rehydration in order to achieve a well hydrated patient at start of surgery.

DETAILED DESCRIPTION:
The patients are not allowed to eat after midnight. Routine premedication is given with paracetamol and oxynorm/oxycontin. Thrombosis and antibiotic prophylaxis is given according to surgical department.

The weight of the patient is notices on the morning of surgery (day 0).

The patient arrives in the morning to the preoperative area. A urinary analysis is taken for urinary colour, creatinine, specific weight, osmolality, microalbuminuria and electrolytes. For 30 patients a volume kinetic analysis of 5 ml/kg infusion of acetated Ringers solution is undertaken between 6.30 and 8.00 am on the morning of surgery. During 15 minutes 5 ml/kg acetated Ringers solution is infused intravenously. Hb is continuously measured noninvasively by Masimo Radical 7 pulse oximeter (MasimoHb) and invasively with maximum 13 samples a 4 ml during 80 minutes (0, 10, 15, 25, 40, 50, 60 and 70 min. Double samples at start and 60 min. The volume kinetic part of the study is finished after 70 min when the patient urinates and the volume is measured.

The patient is taken to the operating theatre and MasimoHb, NT-proBNP, Troponin T hs, pl-lactate, PI och PVI (stable value during 5 min) is registered before anaesthesia. Avoid having blood pressure cuff and pulse oximeter for PVI analysis on the same arm. Aim at PI > 1 to get a reliable registration of PVI, otherwise try another finger.

Anaesthesia: Epidural anaesthesia according to clinical praxis (activated after the first volume optimisation and kept activated during surgery) and anaesthesia according to clinical practise. The ventilation during anaesthesia is maintained using volume controlled mode, tidal volume 7 ml/kg (ideal weight, using the formula: men 50 + 0.91(height in centimetre -152.4); women 45.5 + 0.91(height in centimetre -152.4)), PEEP 5 - 10 cmH2O, respiratory rate to achieve normocapnia. Tidal volume and PEEP is maintained during surgery. The Doppler sond is placed after anaesthesia induction and after that the gastric sond is placed.

During induction of anaesthesia an amount of u to 500 ml colloid solution as well as intermittently ephedrine in small doses of 2.5 - 10 mg can be given for circulatory stability.

Antibiotics are given according to clinical practice.

Preoperative fluid regimen:

Grupp OD:

Basic infusion: Buffered glucose 2.5% 1000 ml 2 ml/kg/h. The first volume optimization of stroke volume (SV) takes place after anaesthesia induction and a stable baseline of measurement is achieved. Note SV (mean value during 1 min), Flow time corrected (FTC), MasimoHb and PVI (mean value during 1 min). The PVI value is only visualised to the research nurse and not to the attending anaesthesiologist. Administer 3 ml/kg (actual weight) maximum 250 ml hydroxyethyl starch during 5 minutes. Wait for 5 minutes. Note SV, FTC, MasimoHb and PVI. If SV increases more than 10 % a new colloid bolus is given. This is repeated in cycles until SV not increases > 10%, or DO2i > 600 ml/min/m2. For every cycle SV, FTC, MasimoHb and PVI are noted. The first optimization is undertaken before start of surgery.

SV, FTC, MasimoHb and PVI are followed during surgery. If SV is reduced > 10% from the value after the last bolus dose a new volume optimization is repeated as described above.

If more than 30 ml/kg hydroxyethyl starch 60 mg/ml is given, colloid solution is changed to albumin 4% or plasma. Bolus doses of albumin 4% and plasma are also 3 ml/kg with a maximum of 250 ml.

Beside infusion of colloids, acetated Ringers solution 0-1000 ml can be given according to the decision from the attending anaesthesiologist.

Blood loss is replaced ml by ml with colloid until Hb 90 g/l (100 if the patient has an ischemic heart disease or any other condition at the discretion from the attending anaesthesiologist). Thereafter replacement is given1:1 using SAG and colloid/albumin/plasma. If blood loss exceeds half the blood volume replacement is given only using SAG/plasma. Thrombocytes are given according to clinical practice.

Any use of inotropic and vasoactive drugs is documented.

At the end of surgery pl-lactate and Hb is measured invasively and non-invasively (HB). Estimated blood loss is registered.

Grupp PVI:

Basic infusion: Buffered glucose 2.5% 1000 ml 2 ml/kg/h.

The first volume optimization of stroke volume (SV) takes place after anaesthesia induction and a stable baseline of measurement is achieved. Note PVI ( mean value during 1 min), MasimoHb, SV (mean value during 1 min) and Flow time corrected (FTC). Data from the oesophagus doppler is only visualised to the research nurse and not to the attending anaesthesiologist. Administer 3 ml/kg (actual weight) maximum 250 ml hydroxyethyl starch during 5 minutes. Wait for 5 minutes. Note SV, FTC, MasimoHb and PVI. If PVI is >10 % and reduced give a new colloid bolus. For every cycle SV, FTC, MasimoHb and PVI are noted. The first optimization is undertaken before start of surgery.

If PVI >10 % the volume optimization is repeated as described above. If more than 30 ml/kg hydroxyethyl starch 60 mg/ml is given, colloid solution is changed to albumin 4% or plasma. Bolus doses of albumin 4% and plasma are also 3 ml/kg with a maximum of 250 ml.

Beside infusion of colloids, acetated Ringers solution 0-1000 ml can be given according to the decision from the attending anaesthesiologist.

Blood loss is replaced ml by ml with colloid until Hb 90 g/l (100 if the patient has an ischemic heart disease or any other condition at the discretion from the attending anaesthesiologist). Thereafter replacement is given1:1 using SAG and colloid/albumin/plasma. If blood loss exceeds half the blood volume replacement is given only using SAG/plasma. Thrombocytes are given according to clinical practice.

Any use of inotropic and vasoactive drugs is documented.

At the end of surgery pl-lactate and Hb is measured invasively and non invasively (HB). Estimated blood loss is registered.

Both groups: If the patients' perioperative course demands that the anaesthesiologists in charge deviate from the study protocol the reason for this is registered in the CRF.

All patients have a urinary bladder catheter or cystofix as decided by the surgeon. The temperature of the patient is measured. Hot air blanked is used to prevent hypothermia.

Post-operatively after 12-24 hours and 36-48 hours pl-NT-proBNP and pl-troponinThs are measured.

The patients weight is registered the morning on the day after surgery (day 1).

Date for end of hospital stay is registered.

A blinded team registers postoperative complications on the 3d day after surgery according to a preset protocol. The record is also reviewed retrospectively to document all complications during the first 30 days after surgery.

For patients 1-75 Doppler and PVI are recorded simultaneously to allow analysis of concordance between PVI and Doppler as guide to fluid optimization. Also biochemical analyses of cardiac enzymes as part of the study are undertaken in patients 1-75. For patients 1-150 the outcome measure postoperative complications is registered.

ELIGIBILITY:
Inclusion Criteria:

1. Open abdominal surgery under general anaesthesia with a planned operation time of at least 120 minutes
2. Age ≥ 18 years

Exclusion Criteria:

1. Anaesthesia risk classification ASA ≥ 4
2. Arrhythmia; atrial fibrillation or multiple extra systoles
3. Aortic - or mitral insufficiency with hemodynamic influence
4. Patients who at the preoperative visit by the responsible anaesthesiologist is planned for a more advanced cardiovascular monitoring. The following monitoring is accepted in the study: invasive blood pressure, 5-lead ECG, central venous pressure and urinary output per hour.
5. Patients with a pulmonary or other disease that prevents ventilation using a tidal volume of 7 ml/kg (ideal weight) or a positive end expiratory pressure of 5 -10 cm H2O
6. Contra indication against synthetic colloids as severely impaired renal or liver function, hyper natremia or allergy to synthetic colloids
7. Laparoscopic surgery
8. Liver surgery
9. Surgery including thoracotomy
10. Contraindications against an oesophageal probe such as severe oesophageal varicose veins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
ml colloid infusion | During surgery (2-8 hours)
  Volume colloid fluid to achieve volume optimisation for guidance using Pleth Variability Index and oesophageal doppler, respectively (comparison between groups)
Correlation between ml colloid infusion and dehydration level | During surgery (2-8 hours)
  Correlation between level of dehydration measured by volume kinetics and urinary analysis, and correlation between these two circumstantials and the volume of colloids given for the first volume optimisation using Pleth Variability Index or oesophageal doppler

SECONDARY OUTCOMES:
Days | Days of hospital stay in connection with surgery, usually 2-10 days
  Length of hospital stay
Complications (number) | Complications occuring up to 30 days after surgery
  Number of complications using a prospective classification
NT-pro-BNP | Measured up to 2 days after surgery
  Cardiac stress measured by NT-pro-BNP

CONTACTS AND LOCATIONS:
Overall Officials: Lena Nilsson, MD PhD, Principal Investigator — Anestesi- och operationskliniken, Universitetssjukuset, SE 58183 Linköping, Sweden
Locations (1):
- Anestesi-och operationskliniken, Linköping, Sweden

REFERENCES:
- [Background] Brandstrup B, Tonnesen H, Beier-Holgersen R, Hjortso E, Ording H, Lindorff-Larsen K, Rasmussen MS, Lanng C, Wallin L, Iversen LH, Gramkow CS, Okholm M, Blemmer T, Svendsen PE, Rottensten HH, Thage B, Riis J, Jeppesen IS, Teilum D, Christensen AM, Graungaard B, Pott F; Danish Study Group on Perioperative Fluid Therapy. Effects of intravenous fluid restriction on postoperative complications: comparison of two perioperative fluid regimens: a randomized assessor-blinded multicenter trial. Ann Surg. 2003 Nov;238(5):641-8. doi: 10.1097/01.sla.0000094387.50865.23. PMID 14578723
- [Background] Abbas SM, Hill AG. Systematic review of the literature for the use of oesophageal Doppler monitor for fluid replacement in major abdominal surgery. Anaesthesia. 2008 Jan;63(1):44-51. doi: 10.1111/j.1365-2044.2007.05233.x. PMID 18086070
- [Background] Cannesson M, Desebbe O, Rosamel P, Delannoy B, Robin J, Bastien O, Lehot JJ. Pleth variability index to monitor the respiratory variations in the pulse oximeter plethysmographic waveform amplitude and predict fluid responsiveness in the operating theatre. Br J Anaesth. 2008 Aug;101(2):200-6. doi: 10.1093/bja/aen133. Epub 2008 Jun 2. PMID 18522935
- [Background] Gan TJ, Soppitt A, Maroof M, el-Moalem H, Robertson KM, Moretti E, Dwane P, Glass PS. Goal-directed intraoperative fluid administration reduces length of hospital stay after major surgery. Anesthesiology. 2002 Oct;97(4):820-6. doi: 10.1097/00000542-200210000-00012. PMID 12357146
- [Background] Svensen CH, Olsson J, Hahn RG. Intravascular fluid administration and hemodynamic performance during open abdominal surgery. Anesth Analg. 2006 Sep;103(3):671-6. doi: 10.1213/01.ane.0000226092.48770.fe. PMID 16931679
- [Derived] Hahn RG. Detection of low urine output by measuring urinary biomarkers. BMC Nutr. 2024 Jan 12;10(1):13. doi: 10.1186/s40795-024-00823-3. PMID 38217039
- [Derived] Hahn RG, Wuethrich PY, Zdolsek JH. Can perioperative hemodilution be monitored with non-invasive measurement of blood hemoglobin? BMC Anesthesiol. 2021 May 6;21(1):138. doi: 10.1186/s12871-021-01351-4. PMID 33957864
- [Derived] Bahlmann H, Hahn RG, Nilsson L. Pleth variability index or stroke volume optimization during open abdominal surgery: a randomized controlled trial. BMC Anesthesiol. 2018 Aug 18;18(1):115. doi: 10.1186/s12871-018-0579-4. PMID 30121072
- [Derived] Hahn RG, Bahlmann H, Nilsson L. Preoperative fluid retention increases blood loss during major open abdominal surgery. Perioper Med (Lond). 2017 Sep 2;6:12. doi: 10.1186/s13741-017-0068-1. eCollection 2017. PMID 28878889
- [Derived] Hahn RG, Bahlmann H, Nilsson L. Dehydration and fluid volume kinetics before major open abdominal surgery. Acta Anaesthesiol Scand. 2014 Nov;58(10):1258-66. doi: 10.1111/aas.12416. PMID 25307711